CLINICAL TRIAL: NCT04639726
Title: A Randomized, Placebo-Controlled, Single-Center, Crossover Study to Evaluate the Effects of Pre-Meal Whey Protein Microgels Administration on Post-Prandial Glycemic Response in Patients with Type 2 Diabetes.
Brief Title: A Study to Evaluate the Effects of Pre-Meal Whey Protein Microgels Administration on Post-Prandial Glycemic Response.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 19.14.CLI
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dietary Supplement
MeSH Terms: interventions — Water; Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whey Protein (Active Comparator)
  Interventions: Dietary Supplement: Whey Protein Micro Gel
- Placebo (Placebo Comparator)
  Interventions: Other: Water without Whey Protein.

INTERVENTIONS:
Dietary Supplement: Whey Protein Micro Gel — The test product is whey protein microgels 10g, reconstituted in 125ml water.
  Arms: Whey Protein
Other: Water without Whey Protein. — A matching placebo (125ml of water without whey protein) will be used as control.
  Arms: Placebo

SUMMARY:
This is a mechanistic, randomized, investigator-blinded, placebo-controlled, single-center, crossover study designed to evaluate the effects of premeal administration of whey protein microgels compared to placebo on postprandial glycemia in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign written informed consent prior to study entry.
* Male or female, >18 years of age.
* Established diagnosis of type 2 diabetes (documented by either HbA1c 6.5 - 10.0% or a history of type 2 diabetes diagnosis).
* Treatment naïve or on active therapy with metformin at a daily dose of 1000-3000mg at screening. Dose of metformin must have been stable for at least 3 months prior to screening.
* Patients must have a hematocrit value greater than or equal to 34.0% for females and 40% for males.
* Patients must have a hemoglobin value greater than or equal to 11.0 g/dL for females and 13.5 g/dL for males.

Exclusion Criteria:

* Fasting plasma glucose >220mg/dl at screening.
* Impaired kidney function, epidermal growth factor receptor of <60mL/min/1.73m2 at screening.
* BMI >40kg/m2.
* Elevated liver transaminase > 3 upper limit of normal at screening.
* Ongoing or recent (i.e. < 3month) treatment with any oral or injectable glucose-lowering drug other than metformin.
* Ongoing or recent (i.e. < 3month) injectable insulin therapy.
* Ongoing or recent (i.e. < 3 month) weight loss interventions (e.g. dietary weight loss programs) or any history of bariatric surgery or any documented weight loss >5% within previous 6 months.
* Ongoing or recent (i.e. < 3 month) treatment with anorectic drugs, systemic steroids, medications known to affect gastric motility, or any condition known to affect gastro-intestinal integrity and food absorption.
* Major medical/surgical event requiring hospitalization in the last 3 months.
* Known allergy and intolerance to product components or acetaminophen.
* Alcohol intake higher than 2 servings per day. A serving is 0.4dl of strong alcohols, 1dl of red or white wine, or 3dl of beer.
* Are unable to comply with protocol procedures in the opinion of the investigator.
* Have a hierarchical link with the research team members.
* Positive pregnancy test at screening.
* Patients who have been dosed in another clinical trial with any investigational drug/new chemical entity within 30 days or 5 half-lives (whichever is longer) prior to screening, or patients currently participating in any investigational trial.
* Donation of blood or significant amount of blood loss within 8 weeks prior to screening. Patients must also agree to not donate blood within 8 weeks after their last visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Post-prandial glycemic excursion. | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Incremental area under the curve post-prandial glycemic excursion (iAUC 0-3 hours)

SECONDARY OUTCOMES:
2h post-prandial glucose | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Incremental area under the curve 2hours post-prandial glucose levels
Total glucose | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Total glucose AUC (tAUC 0-3hours)
Plasma glucose | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Plasma glucose iCmax
Plasma glucose | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Plasma glucose Tmax
Plasma glucose | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Plasma glucose AUC (iAUC 0-4hours, tAUC 0-4hours)
Serum insulin | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Serum insulin (iAUC 0-3hours, iCmax, Tmax, tAUC 0-3hours)
Plasma glucagon | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Plasma glucagon (iAUC 0-3hours, iCmax, Tmax, tAUC 0-3hours)
Plasma Glucagon-like Peptide-1 | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Plasma GLP-1 (iAUC 0-2hours, iCmax, Tmax, tAUC 0-2hours)
Plasma Gastric Inhibitory Polypeptide | -15, 0, 30, 60, 90, and 120 minutes.
  Plasma GIP (iAUC 0-2hours, iCmax, Tmax, tAUC 0-2hours)
Plasma ghrelin | -15, 0, 30, 60, 90, and 120 minutes.
  Plasma ghrelin (iAUC 0-2hours, iCmax, Tmax, tAUC 0-2hours)
Plasma cholecystokinin | -15, 0, 30, 60, 90, and 120 minutes.
  Plasma cholecystokinin (CCK) (iAUC 0-2hours, iCmax, Tmax, tAUC 0-2hours)
Plasma peptide | -15, 0, 30, 60, 90, and 120 minutes.
  Plasma peptide-YY (PYY) (iAUC 0-2hours, iCmax, Tmax, tAUC 0-2hours)
Serum triglycerides | -15, 0, 30, 60, 90, and 120 minutes.
  Serum triglycerides (iAUC 0-2hours, iCmax, Tmax, tAUC 0-2hours)
Gastric emptying | -15, 0, 15, 30, 45, 60, 90, 120, 180, and 240 minutes.
  Gastric emptying (AUC 0-4hours, Cmax and Tmax for acetaminophen)
Beta-cell function I | -15, 0, 30, 60, 90, and 120 minutes.
  Beta-cell function I: AUC insulin 0-3hours: AUC glucose 0-3hours ratio
Beta-cell function II | -15, 0, 30, 60, 90, and 120 minutes.
  Beta-cell function II: Insulinogenic index (IGI): [insulin (30-0 minutes) (μU/mL)/glucose (30-0 minutes) (mg/dL)]

OTHER OUTCOMES:
Plasma glucose | 0, 15, 30, 45, 60, 90, 120, 150, 180, and 240 minutes
  Plasma glucose at individual timepoints
Serum insulin | 0, 15, 30, 45, 60, 90, 120, 150, 180, and 240 minutes
  Serum insulin at individual timepoints
Plasma glucagon | 0, 15, 30, 45, 60, 90, 120, 150, 180, and 240 minutes)
  Plasma glucagon at individual timepoints
Plasma glucose | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Plasma glucose (iAUC 0-2hours, iAUC 0-1hour, tAUC 0-2hours, tAUC 0-1hour)
Serum insulin | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Serum insulin (iAUC 0-4hours, tAUC 0-4hours, iAUC 0-2hours, tAUC 0-2hours, iAUC 0-1hour, tAUC 0-1hour)
Plasma glucagon | -30, -15, 0, 15, 30, 45, 60, 120,150, 180, and 240 minutes.
  Plasma glucagon (iAUC 0-4hours, tAUC 0-4hours, iAUC 0-2hours, tAUC 0-2hours, iAUC 0-1hour, tAUC 0-1hour)
Plasma GLP-1 | -15, 0, 30, 60, 90, 120 minutes.
  Plasma GLP-1 (iAUC 0-1hour, tAUC 0-1hour)
Plasma GIP | -15, 0, 30, 60, 90, 120 minutes.
  Plasma GIP (iAUC 0-1hour, tAUC 0-1hour)
Serum triglycerides | -15, 0, 30, 60, 90, 120 minutes
  Serum triglycerides (iAUC 0-1hour, tAUC 0-1hour)
Plasma ghrelin | -15, 0, 30, 60, 90, 120 minutes
  Plasma ghrelin (iAUC 0-1hour, tAUC 0-1hour)
Plasma cholecystokinin | -15, 0, 30, 60, 90, 120 minutes
  Plasma cholecystokinin (CCK) (iAUC 0-1hour, tAUC 0-1hour)
Plasma peptide | -15, 0, 30, 60, 90, 120 minutes.
  Plasma peptide-YY (PYY) (iAUC 0-1hour, tAUC 0-1hour)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No